CLINICAL TRIAL: NCT03366948
Title: Internet Gaming Disorder Prevalence of Teenager Psychiatric Inpatient of 4 Psychiatric Units of French Region Auvergne-Rhône-Alpes
Brief Title: Internet Gaming Disorder and Psychiatric Disorder
Acronym: IGDPD
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL17_0685
Record Dates: First submitted 2017-12-04; First posted 2017-12-08 (Actual); Last update posted 2019-08-13 (Actual); Status verified 2019-08

CONDITIONS: Psychiatric Disorder
MeSH Terms: conditions — Mental Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: IGDT-10 self-administered questionnaire — Patients and their parents will answer the French version of the IGDT-10 self-administered questionnaire (IGDT-10-P in the parents 'questionnaire).
  The IGDT-10 is a self-administered questionnaire based on DSM-5 internet gaming disorder criteria and the IGDT-10-P is a parental version specially adapted from the IGDT-10 for this study.

SUMMARY:
The fifth edition of the Diagnostic and Statistical Manual of Mental Disorders (DSM-5) recently identified Internet gaming disorder as a new potential psychiatric disorder which need further research. Several studies showed the important prevalence of psychiatric disorders among patients suffering from internet gaming disorder. Investigators hypothesize that on an other side the prevalence of internet gaming disorder among patients suffering from psychiatric disorders shall be high but it has never been studied yet.

The main goal of this trial is to examine the prevalence of internet gaming disorder using the Internet Gaming Disorder Test-10 (IGDT-10) among inpatient aged from 12 to 17 of 4 psychiatric units of French region Auvergne-Rhône-Alpes.

Secondary goals will be to assess a parental version of the IGDT-10 (IGDT-10-P) and to compare the two versions.

IGDT-10 will be passed during 6 months to every inpatient and IGDT-10-P to their parents within the 21 first days of the hospitalisation.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged from 12 to 17
* Parents of the patient, older than 18 years old
* Patients hospitalized in 4 psychiatric units of French region Auvergne-Rhône-Alpes

Exclusion Criteria:

* Patient and/or theirs parents are not fluent in French
* Intellectual deficit (known intelligence quotient below 70)
* Behaviour disorder making impossible to pass the questionnaire

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Patient aged from 12 to 17 of 4 psychiatric units of French region Auvergne-Rhône-Alpes and their parents.
Sampling Method: Non-Probability Sample
Enrollment: 102 (Actual)
Dates: Start 2018-03-16 (Actual); Primary Completion 2018-09-14 (Actual); Study Completion 2018-09-14 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with a IGDT-10 score above 5 | In the first 21 days after the admission in the psychiatric unit.
  The 10-item Internet Gaming Disorder is a 10 dichotomous items self-assessment scale corresponding to the 9 diagnostic criteria of the DSM-5 IGD (the last item is split in two but should only be counted once). In agreement with DSM-5, a diagnosis of IGD is considered positive if 5 criteria are validated. Each criterion is filled by the patient as "never", "sometimes" or "often", a criterion is validated if it is reported to be present "often" in the last 12 months according to DSM-5 guidelines. The Ten-Item Internet Gaming Disorder Test (IGDT-10) by Király et al. was validated in English for a population of 14 to 64 years10 then in French in adults by Laconi et al.29. This is a valid and reliable scale.

CONTACTS AND LOCATIONS:
Locations (5):
- France (5):
  - Service de pédopsychiatrie Centre hospitalier Pierre Oudot, Bourgoin
  - Psychopathologie du Développement Hôpital Femme Mère Enfant, Bron
  - Service de psychiatrie adulte Hôpital Pierre Wertheimer-GHE, Bron
  - Service de pédopsychiatrie - Unité H.Flavigny Centre hospitaliser Le Vinatier, Bron
  - Service de pédopsychiatrie - Unité Adolescents ULYSSE - Centre hospitalier St Jean-de-Dieu, Lyon

IPD SHARING:
Plan to Share IPD: No